CLINICAL TRIAL: NCT03948841
Title: Measurement Variability of Liver Metastases From Neuroendocrine Tumors on Different Magnetic Resonance Imaging Sequences
Acronym: NETMRI
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2018Ao006
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine tumor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuroendocrine tumor: Patients with liver metastasis from neuroendocrine tumor
  Interventions: Other: magnetic resonance imaging

INTERVENTIONS:
Other: magnetic resonance imaging

SUMMARY:
The aim of our study is to assess variability of measurements of liver metastases from neuroendocrine tumors (NET) on different magnetic resonance imaging (MRI) sequences.

In this institutional review board-approved retrospective study from January 2011 to December 2012, all liver MRIs performed at our department in patients with proven liver metastases from NETs and with at least one measurable lesion according to Response evaluation criteria in solid tumors (RECIST 1.1) were included.

DETAILED DESCRIPTION:
The aim of our study is to assess variability of measurements of liver metastases from neuroendocrine tumors (NET) on different magnetic resonance imaging (MRI) sequences.

In this institutional review board-approved retrospective study from January 2011 to December 2012, all liver MRIs performed at our department in patients with proven liver metastases from NETs and with at least one measurable lesion according to Response evaluation criteria in solid tumors (RECIST 1.1) were included. Up to two lesions were selected by an independent radiologist on T2-weighted images and marked by an arrow. Three reviewers (attending radiologist R1, fellow R2, senior R3) independently obtained long axis measurements of 135 metastases in 30 patients, on T2, diffusion-weighted imaging (DWI) with three b values (50, 400, 800), arterial, portal and late phases after gadolinium ), and during two distant separate sessions. Intraclass correlation coefficients and Bland-Altman plots were used to assess intra-and interobserver variability.

ELIGIBILITY:
inclusion criteria :

* Patients with liver metastasis from neuroendocrine tumor
* Patients with a magnetic resonance imaging in Reims university hospital
* Patients with at least one measurable lesion according to Response evaluation criteria in solid tumors

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver metastasis from neuroendocrine tumor with a magnetic resonance imaging in Reims university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
variability of measurements of liver metastases from neuroendocrine tumors (NET) on different magnetic resonance imaging (MRI) sequences. | Day 0
  calculation of intraclass correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Lestra T, Kanagaratnam L, Mule S, Janvier A, Brixi H, Cadiot G, Dohan A, Hoeffel C. Measurement variability of liver metastases from neuroendocrine tumors on different magnetic resonance imaging sequences. Diagn Interv Imaging. 2018 Feb;99(2):73-81. doi: 10.1016/j.diii.2017.12.009. Epub 2018 Jan 12. PMID 29339222